CLINICAL TRIAL: NCT05700110
Title: Porto-venous Radiomics in Pancreatic Cancer: A Multi-centre Retrospective Cohort Study Investigating the Use of Pre-operative CT Radiomic Features to Predict Surgical Resection Margin in Pancreatic Head Malignancy
Brief Title: Porto-Venous Radiomics in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5615
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-Interventional — Non-interventional

SUMMARY:
Multi-centre Retrospective Observational Cohort study of patients who underwent pancreaticoduodenectomy from 01/01/2005 to 01/02/2022 with histologically confirmed pancreatic head malignancy

DETAILED DESCRIPTION:
Pancreatic cancers are often inoperable at diagnosis, with only 13-22% of patients being suitable for surgical resection.1 Surgery is the only curative therapeutic option for pancreatic cancer and higher rates of long-term patient survival following surgery are seen in patients where the tumour is completely removed (termed R0 resection). However a majority of those patients who undergo surgery will develop tumour recurrence at the primary surgical site or a distant location. The likelihood of cancer recurrence following surgery increases when there is involvement of major blood vessels that lie adjacent to the pancreas. This involvement is often microscopic in nature and only detected after surgery when the surgical specimen is examined microscopically (termed R1 resection). Pre-operative cross-sectional imaging (usually Computed Tomography (CT) is the standard tool used to assess the risk of R1 resection prior to pancreatic cancer. However this approach significantly overestimates the number of patients with a resectable tumour as a significant proportion ultimately have an R1 resection after surgery. If there is felt to be an increased risk of R1 resection prior to surgery the patient can be offered oncological treatment prior to surgery to improve the rates of R0 resection that in turn improve long-term patient survival.

The emerging field of Radiomics offers the opportunity to stratify patients undergoing pancreatic cancer surgery into those at risk of R1 resection prior to surgery. Radiomics has emerged as a valuable adjunct to medical decision making over the past 10 years. The basic premise is to extract and analyse large amounts of information not usually visible to the human eye from medical images, and it is increasingly being used in the field of cancer diagnostics. The aim of this study is to employ 3D radiomic analyses to pre-operative CT scan images for cases of pancreatic head cancer that underwent surgical resection, to determine whether this information could be used to predict R0 and R1 resection margins pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pancreaticoduodenectomy/Whipple's surgery for pancreatic head malignancy between 01/01/2005 and 01/02/2022.
* Pre-operative Computed Tomographic images within 90 days prior to surgical resection.
* Post-operative histological confirmation of pancreatic ductal adenocarcinoma (PDAC), ampullary adenocarcinoma (AA), distal bile duct carcinoma (DBC), pancreatic neuroendocrine tumours (NET/NEC), duodenal adenocarcinoma (DA) or duodenal gastro-intestinal stromal tumours (GIST).

Exclusion Criteria:

* Postoperative surgical histology confirming benign pathology, metastatic disease or invasive malignancy arising from sites other than duodenum, pancreatic head or distal common bile duct.
* Patients who underwent distal pancreatectomy or total pancreatectomy as their primary surgical procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients on locally maintained patient databases recorded as having undergone a pancreaticoduodenectomy or Whipple's surgery on or after 01/01/2005 will be screened by the local clinical team for eligibility.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-05-05 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
To develop a Radiomics model based on pre-operative CT porto-venous phase imaging that accurately predicts Resection Margin status in pancreatic head malignancy | 12 months from recruitment of first patient
  R classification of resection margin status on post-operative histological analysis as per the Royal College of Pathologists classification

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No